CLINICAL TRIAL: NCT06904300
Title: A Randomized, Controlled, Multi-center Phase II Study of Ivonescimab (AK112) Plus Paclitaxel Versus Paclitaxel With or Without Ramucirumab as Second-line Therapy in Subjects With Advanced Gastric or Gastroesophageal Junction（G.GEJ）Cancer Who Failed Immunochemotherapy
Brief Title: Ivonescimab (AK112) Plus Paclitaxel as Second-line Therapy in Patients With Advanced G/GEJ Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Feng Wang, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AK112-IIT-003
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Gastric (Cardia, Body) Cancer
Keywords: immunotherapy
MeSH Terms: conditions — Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): AK112 (20 mg/kg IV, D1/D15) + paclitaxel (80 mg/m² IV, D1/D8/D15), Q4W
  Interventions: Drug: AK112 + paclitaxel
- Group B (Active Comparator): Paclitaxel (80 mg/m² IV, D1/D8/D15) ± ramucirumab (8 mg/kg IV, D1/D15), Q4W
  Interventions: Drug: Paclitaxel ± ramucirumab

INTERVENTIONS:
Drug: AK112 + paclitaxel — AK112 (20 mg/kg IV, D1/D15) + paclitaxel (80 mg/m² IV, D1/D8/D15), Q4W
  Arms: Group A
Drug: Paclitaxel ± ramucirumab — Paclitaxel (80 mg/m² IV, D1/D8/D15) ± ramucirumab (8 mg/kg IV, D1/D15), Q4W
  Arms: Group B

SUMMARY:
A Randomized, Controlled, Multi-center Phase II Study of Ivonescimab (AK112) plus Paclitaxel versus Paclitaxel with or without Ramucirumab as second-line therapy in subjects with advanced gastric or gastroesophageal junction（G/GEJ）cancer who failed immunochemotherapy

DETAILED DESCRIPTION:
This is a randomized, controlled, multi-center Phase II trial (N ≈ 110) conducted in China to assess the safety and antitumor activity of AK112 combined with paclitaxel versus paclitaxel with or without ramucirumab in subjects with advanced gastric/gastroesophageal junction adenocarcinoma who failed immunochemotherapy. The study objective was to assess the progression-free survival (PFS) of AK112 combined with paclitaxel versus paclitaxel with or without ramucirumab in subjects with advanced gastric/gastroesophageal junction adenocarcinoma who failed immunochemotherapy. The primary endpoint was PFS assessed by RECIST v1.1, and the secondary endpoints were ORR, OS, DoR, time to response (TTR), DCR, and incidence/severity of adverse events (AEs) graded by NCI CTCAE v5.0. Eligible patients with progression after PD-1/L1 inhibitor plus platinum chemotherapy will be stratified by peritoneal metastasis (present vs. absent) and randomized 1:1 to: Group A (n=55): AK112 (20 mg/kg IV, D1/D15) + paclitaxel (80 mg/m² IV, D1/D8/D15), Q4W; Group B (n=55): Paclitaxel (80 mg/m² IV, D1/D8/D15) ± ramucirumab (8 mg/kg IV, D1/D15), Q4W. Treatment continues until disease progression, intolerable toxicity, or investigator-determined clinical futility.Tumor assessments occur every 8 weeks (±7 days) via RECIST v1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent provided
2. Age ≥18 and ≤75 years, regardless of gender
3. Histologically or cytologically confirmed advanced or metastatic gastric adenocarcinoma or gastroesophageal junction adenocarcinoma
4. Prior treatment failure with PD-1/L1 inhibitor combined with platinum-based chemotherapy; no other systemic antitumor therapy allowed (only first-line therapy permitted, with initial immunotherapy duration ≥12 weeks).Note: Patients who previously received adjuvant/neoadjuvant PD-1 inhibitor plus platinum-based chemotherapy for non-metastatic disease or curative-intent platinum chemoradiotherapy + PD-1 inhibitor for locally advanced or recurrent/metastatic disease are eligible if disease progression occurred within <6 months after the last treatment and no subsequent systemic therapy was administered.
5. ECOG performance status of 0-1
6. Life expectancy ≥3 months
7. At least one measurable lesion per RECIST v1.1. Previously irradiated lesions may qualify as target lesions if evidence of post-radiotherapy progression exists and no alternative target lesions are available.
8. Adequate organ function:

   Hematology (without transfusions/growth factors for 7 days): ANC ≥1.5×10⁹/L; platelets ≥100×10⁹/L; hemoglobin ≥90 g/L.

   Liver: Total bilirubin ≤1.5×ULN; AST/ALT ≤2.5×ULN (≤5×ULN for hepatic metastases); albumin ≥28 g/L.

   Kidney: Serum creatinine ≤1.5×ULN and CrCl ≥50 mL/min; urine protein <2+ or 24-hour urinary protein <1.0 g.

   Coagulation: INR/PT ≤1.5×ULN (unless on anticoagulants with therapeutic ranges maintained).

   Cardiac: LVEF ≥50%.
9. For females of childbearing potential: Negative pregnancy test within 3 days prior to treatment; highly effective contraception required during screening and for 120 days post-treatment. Postmenopausal women (amenorrhea ≥1 year) or surgically sterilized females are exempt.
10. For non-sterilized males with childbearing partners: Effective contraception during screening and for 120 days post-treatment.
11. Willingness and ability to comply with protocol-specified visits, treatments, and laboratory tests.

Exclusion Criteria:

1. Histologically or cytologically confirmed as other pathological types (e.g., squamous cell carcinoma, undifferentiated carcinoma, neuroendocrine carcinoma). Mixed pathological types will be categorized based on the predominant component; only subjects with >70% adenocarcinoma component confirmed by a pathologist may enroll.
2. History of other malignancies within 3 years prior to enrollment. Exceptions include malignancies cured by local therapy (e.g., basal or squamous cell skin cancer, superficial bladder cancer, in situ cervical or breast cancer).
3. Systemic anti-cancer therapy (e.g., chemotherapy, radiotherapy, immunotherapy, targeted therapy [<2 weeks for small-molecule agents], biologics) within 3 weeks prior to first dose; palliative local therapy for non-target lesions within 2 weeks.
4. Prior immunotherapy other than PD-1/PD-L1 inhibitors, including checkpoint inhibitors (anti-CTLA-4, anti-CD47, anti-SIRPα, anti-LAG-3), checkpoint agonists (ICOS, CD40, CD137, GITR, OX40), cell therapies, or biologics targeting tumor immunity.
5. Prior treatment with ramucirumab, VEGFR2 antagonists, or other VEGFR2-targeting antibodies/proteins.
6. Prior use of taxane-based agents (e.g., paclitaxel, docetaxel) in first-line systemic therapy.
7. Prior PD-1/PD-L1 inhibitor treatment with any of the following:

   1. Grade ≥3 irAEs (excluding endocrine irAEs), irAEs leading to permanent discontinuation, Grade 2 immune-related cardiotoxicity, or any-grade neurological/ocular irAEs.
   2. Unresolved toxicities from prior PD-1/PD-L1 therapy (not resolved to ≤Grade 1). Grade ≥2 endocrine toxicities are allowed if stable and asymptomatic under replacement therapy.
   3. IrAEs requiring non-corticosteroid immunosuppressants or recurrent irAEs necessitating systemic corticosteroids.
8. Hypersensitivity to any study drug component or history of severe allergic reactions to monoclonal antibodies.
9. Bleeding diathesis or coagulation disorders.
10. Imaging showing tumor invasion of adjacent organs/vessels, necrosis, or cavitation posing risk of perforation/hemorrhage.
11. Major surgery/trauma within 30 days prior to first dose or planned surgery within 30 days post-dose; minor surgery within 3 days prior to first dose (excluding PICC/port placement).
12. Gastrointestinal risks:Esophagogastric varices, severe ulcers, unhealed wounds, perforation, fistula, abscess, or acute bleeding within 6 months; Arterial thromboembolism or Grade ≥3 venous thromboembolism (per NCI CTCAE v5.0), TIA, stroke, hypertensive crisis, or COPD exacerbation within 6 months; Uncontrolled hypertension (≥160/100 mmHg on oral therapy).
13. Cardiac history:Myocarditis, cardiomyopathy, malignant arrhythmia; Unstable angina, MI, NYHA Class ≥2 heart failure, or aortic aneurysm within 12 months; Poorly controlled arrhythmias or ischemia.
14. Active autoimmune disease requiring systemic treatment within 2 years (excluding hormone replacement).
15. Symptomatic effusions requiring diuretics or drainage (pleural, pericardial, or ascites).
16. Severe infection (hospitalization-required/sepsis) within 4 weeks; active infection requiring systemic antibiotics within 2 weeks (excluding antiviral therapy for HBV/HCV).
17. Active tuberculosis (must be ruled out if suspected) or active syphilis.
18. Organ or stem cell transplant history (excluding corneal transplants).
19. Immunodeficiency:HIV-positive; Chronic systemic corticosteroids/immunosuppressants.
20. Chronic viral hepatitis:Active HBV (HBsAg-positive with HBV DNA >500 IU/mL or >2500 copies/mL); Active HCV (allowed if cured or HCV RNA-negative).
21. Live/attenuated vaccines administered within 30 days prior to first dose or planned during the study (inactivated vaccines permitted).
22. Pregnancy, lactation.
23. History of psychiatric disorders, substance abuse, or alcoholism.
24. Other conditions deemed ineligible by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 12-24 months

SECONDARY OUTCOMES:
ORR | 12-24 months
DCR | 12-24 months
DoR | 12-24 months
OS | 12-24 months